CLINICAL TRIAL: NCT00731926
Title: Effect of Antioxidant on Endurance Performance in Healthy Men -Double Blind Randomized Placebo and Active Controlled Trial-
Brief Title: Effect of Antioxidant on Endurance Performance in Healthy Men
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: University of California, Davis (Other)
Responsible Party: Sang-chul Lee MD., Ph.D / chief director, Institute of Complementary Alternative Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-0707-028-212
Record Dates: First submitted 2008-05-20; First posted 2008-08-11 (Estimated); Last update posted 2008-08-12 (Estimated); Status verified 2008-08

CONDITIONS: Exercise Tolerance
MeSH Terms: interventions — oligonol; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Dietary Supplement: Oligomerized litchi fruit extract
- 2 (Active Comparator)
  Interventions: Dietary Supplement: VItamin C + Vitamin E mixture
- 3 (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: Oligomerized litchi fruit extract — 100mg at once twice a day for 1 month
  Other Names: oligonol; brand name of oligomerized litchi fruit extract
  Arms: 1
Dietary Supplement: VItamin C + Vitamin E mixture — Vitamin C 400mg + Vitamin E 160IU at once twice a day for 1 month
  Arms: 2
Other: placebo — twice a day for 1 month
  Arms: 3

SUMMARY:
oligomerized litchi fruit extract may enhance the submaximal endurance exercise performance

DETAILED DESCRIPTION:
Regular physical exercise has many beneficial effects, but it has been reported that strenuous exercise could elevate the production of free radical and other reactive oxygen species (ROS) which eventually injure the tissues and decrease the muscle function.So many kinds of antioxidant supplementations have been tried to decrease the muscle fatigue and enhance the exercise performance. polyphenolic flavonoids abundant in fruits and leafy vegetables have strong antioxidant effect. oligomerized litchi fruit extract has strong antioxidant capacity and higher bioavailability compared to that of grape seed polyphenol. The aim of this study was to determine whether oligomerized litchi fruit extract could induce endurance exercise performance more than Vit C + Vit E mixture or placebo could do. Therefore, we designed double blind randomized controlled trial, setting the change of running time to exhaustion under submaximal treadmill test as the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* healthy men over 20 years old non-smoker

Exclusion Criteria:

* BMI>25 or body fat>25% he who intakes the antioxidant supplement in recent 2 weeks

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2007-09; Primary Completion 2008-01 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
change of running time to exhaustion under 80% of maximal heart rate | 1 month

SECONDARY OUTCOMES:
VO2max, anaerobic threshold | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Sang-chul Lee, professor, Principal Investigator — Institute of Complementary Alternative Medicine SNUMC